CLINICAL TRIAL: NCT05139108
Title: The Association Between Transesophageal Echocardiography Monitoring and the Incidence of Postoperative Acute Kidney Injury in Coronary Artery Bypass Grafting：a Prospective Observational Study
Brief Title: TEE Monitoring and the Incidence of Postoperative Acute Kidney Injury in Coronary Artery Bypass Grafting
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Collaborators: Zibo Central Hospital (Other Government)
Responsible Party: Principal Investigator, Lili Cao, professor, Qianfoshan Hospital
Other Study IDs: QianfoshanH TEE-AKI
Record Dates: First submitted 2021-11-12; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Coronary Artery Bypass Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
TEE has a definite effect on the evaluation of cardiac structure and function in perioperative cardiac surgery. However, in CABG, previous studies on TEE mainly focused on whether to change the surgical plan rather than improve the clinical prognosis. There are few related studies on the evaluation of prognosis, and these studies have low efficacy and inconsistent conclusions. Acute kidney injury is the most common complication of CABG surgery and is independently associated with hospitalization and long-term mortality. In CABG patients, acute kidney injury, in addition to operation-related factors, is closely related to renal perfusion. These patients often exist serious coronary multivessel lesions and right heart dysfunction, which can cause the system obstacle of regurgitation of the inferior vena cava and kidney blood stasis, while the inappropriate rehydration fluid overload will affect kidney blood perfusion, which may be one of the reasons for the kidney injury. Therefore, appropriate volume status plays an important role in maintaining right heart function and renal perfusion. What indicators can the investigators use to effectively evaluate the patient's volume status and monitor the patient's right heart function?

In recent years, ultrasound has been used as an effective tool to assess patient volume status , right heart function, and to guide patient fluid management. Many studies have confirmed that the respiratory variability of inferior vena cava diameter (ΔIVC) measured by TTE has a good correlation with the volume status of patients on mechanical ventilation, which has a high diagnostic value for predicting the fluid responsiveness and guiding fluid management.However, no study has been reported using TEE measurements of ΔIVC to assess volume status and guide fluid management in patients undergoing cardiac bypass surgery. Previous studies have confirmed that TAPSE measured by TTE is independently associated with AKI in ICU patients and can predict the occurrence of AKI in such patients. However, TAPSE monitored by TEE have not been reported in this regard. Can ΔIVC and TAPSE predict the incidence of AKI and major cardiovascular and cerebrovascular adverse events in CABG patients?

Therefore, the investigators designed this observational study to further scientifically confirm the validity and guiding significance of ΔIVC and TAPSE in CABG, so as to protect and improve patients' renal function , reduce postoperative mortality and improve the clinical prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years；
* Patients undergoing elective isolated coronary artery bypass surgery (with or without bypass)；
* In line with ethics, the patients volunteered to take the test and signed the informed consent for the clinical study;

Exclusion Criteria:

* Patients with severe renal insufficiency before surgery;
* Preoperative patients with moderate or more than moderate valvular lesions required surgery;
* Diabetic patients with a history of serious diabetic complications (diabetic ketoacidosis, hyperosmolar coma, various infections, macrovascular lesions, diabetic nephropathy)；
* Patients with TEE contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective coronary artery bypass surgery alone aged ≥18 years in Tertiary hospitals
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
the incidence of postoperative acute kidney injury | Within 7 days after surgery
  acute kidney injury after cardiac surgery

SECONDARY OUTCOMES:
the incidence of major postoperative cardiovascular and cerebrovascular adverse events | Within 30 days after surgery
  major postoperative cardiovascular and cerebrovascular adverse events after cardiac surgery
the incidence of pulmonary complications | Within 30 days after surgery
  pulmonary complications included pulmonary infection,pulmonary atelectasis, acute lung injury, respiratory failure after cardiac surgery
ICU endotracheal intubation time | Within 30 days after surgery
  ICU endotracheal intubation time

CONTACTS AND LOCATIONS:
Overall Officials: yuelan Wang, PH.D, Study Director — Qianfoshan Hospital
Locations (1):
- Shandong Provincial Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu B, Lv M, Wang H, Sun Y, Song X, Dong L, Feng H, Wang Y. Association between transoesophageal echocardiography monitoring indicators and the incidence of postoperative acute kidney injury in coronary artery bypass grafting: a study protocol for a prospective multicenter cohort study. BMJ Open. 2022 Aug 5;12(8):e059644. doi: 10.1136/bmjopen-2021-059644. PMID 36129681